CLINICAL TRIAL: NCT03709004
Title: Effect of Hospital Pacifier Distribution on Breastfeeding Among Mothers at High Risk for Postpartum Depression
Brief Title: Pacifiers and Breastfeeding Among Mothers at Risk for Postpartum Depression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was not funded and is not going to be done.
Sponsor: University of California, Davis (Other)
Collaborators: Benedictine University (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1132743
Record Dates: First submitted 2018-07-17; First posted 2018-10-17 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Breastfeeding; Postpartum Depression
Keywords: Pacifier
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum | interventions — Pacifiers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pacifier (Experimental): Mother given a pacifier during birth hospitalization, along with other baby items
  Interventions: Other: Pacifier
- Control (No Intervention): Mother not given a pacifier, just the other baby items

INTERVENTIONS:
Other: Pacifier — Pacifier given to mom.
  Arms: Pacifier

SUMMARY:
We will enroll 40 mother-infant dyads in a randomized trial exploring the effect of distribution of pacifiers during the birth hospitalization to mothers at high risk for postpartum depression on pacifier use, infant feeding, and maternal stress.

DETAILED DESCRIPTION:
This study is a pilot a randomized controlled trial to determine if pacifier distribution affects breastfeeding among mothers at high risk for postpartum depression. We will recruit 40 mothers of healthy singleton births in a U.S. hospital who are at high risk of postpartum depression and randomly assign them to receive a pacifier or not. We will ascertain pacifier use, maternal stress, and infant feeding behaviors with web-based surveys at 2, 4, 6, 12, 18, and 24 weeks. Mothers will also wear a wristband to detect maternal heart rate variability throughout the first 6 weeks as a marker of maternal stress.

ELIGIBILITY:
Inclusion Criteria:

* Breastfeeding mother/infant dyad, receiving postpartum care at UC Davis Medical Center, maternal personal or family history of depression or postpartum depression, mother 18-45 years of age, infant 12-72 hours of age

Exclusion Criteria:

* infant without congenital anomalies that could affect feeding (cleft lip/palate, chromosomal anomaly, micro or retrognathia), infant preterm (born prior to 37 weeks' gestation), mother unable to participate in English, infant admitted to the neonatal intensive care unit, No smart phone

Ages: 12 Hours to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Infant Feeding - Breastfeeding Status | up to 24 weeks
  Mode of infant feeding: yes or no
Infant Feeding - Breastfeeding Duration | up to 24 weeks
  Breastfeeding duration overall (number of weeks mothers breastfed exclusively and at all)

SECONDARY OUTCOMES:
Pacifier Use | 2, 4, and 6 weeks
  Any use and frequency in the last 24 hours (7-point Likert scale)

OTHER OUTCOMES:
Maternal Stress | 2, 4, 6, 12, 18, and 24 weeks
  Via Perceived Stress Scale (10 items, 5-point Likert scale)
Infant Feeding Efficiency | 2 and 6 weeks
  Volume of breast milk or formula consumed via bottle within the first three minutes of feeding (mL/min); considered in the context of the infants' state (e.g., alert/awake, drowsy) and nipple size

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No